CLINICAL TRIAL: NCT03755674
Title: Influence of Chronobiological and Neuroendocrine Factors in Appetite Regulation and Obesity Treatment
Brief Title: CHRONOtype-adjusted DIET on Weight Loss
Acronym: CHRONO-DIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Juan Jose Hernández Morante, Principal Investigator of Eating Disorders Research Unit, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMAFI14/12-1
Record Dates: First submitted 2018-07-19; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Obesity
Keywords: Obesity; Appetite regulation; Chronotype; Diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHRONOTYPE-ADJUSTED DIET (Experimental): Patients that undergo a chronotype adjusted diet
  Interventions: Procedure: CHRONOTYPE-ADJUSTED DIET
- CONTROL (No Intervention): Patients following a traditional or conventional hypocaloric diet

INTERVENTIONS:
Procedure: CHRONOTYPE-ADJUSTED DIET — Those patients followed a daily caloric distribution attending to their chronotype. In this regards, 'morning' subjects ate a higher quantity of calories at the first part of the day, while 'evening' subjects ate a higher amount of calories at the second half of the day.
  Arms: CHRONOTYPE-ADJUSTED DIET

SUMMARY:
BACKGROUND: Several reports have observed that the alteration of normal biological rhythms is associated with obesity development. In this regard, those subject with the preference for evening seems to be prone to develop obesity. However, the current treatment of obesity does not take into account these aspects OBJECTIVE: To evaluate whether a diet adjusted to patient's chronotype is more effective than the current dietary recommendations.

SUBJECTS/METHODS: 209 subjects take part in a randomized, double-blind clinical trial. 104 subjects followed a typical hypocaloric dietary treatment (CONTROL) and the other 105 subjects undergone a diet with a daily caloric distribution adjusted to their chronotype (CHRONO).

CONCLUSIONS: A chronotype-adjusted diet may be a promising alternative to the classical hypocaloric dietary treatment since the investigator's data indicate a higher effectiveness regarding weight loss when the diet was adjusted to the patient's chronotype.

ELIGIBILITY:
Inclusion Criteria:

* students or staff of the Catholic University of Murcia (UCAM), with an age ranged between 18 and 65 years old

Exclusion Criteria:

* clinically significant illnesses (including type 2 diabetes, chronic heart failure, hepatitis and cancer)
* those taking any medications known to affect body weight (thyroid hormones, corticosteroids, etc.)
* women in special physiological situations (pregnant, lactating).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Total weight loss, in percentage, from baseline to end-of-treatment | 12 weeks
  Percentage of weight loss, measured with a scale, from baseline weight (100% body weight) since body weight after 12 weeks of treatment (final body weight). Percentage of body weight was then measured as Total Weight Loss (%) = (Final body weight - Baseline body weight) / baseline body weight x 100.

SECONDARY OUTCOMES:
BMI loss | 12 weeks
  BMI decrease from baseline
Anthropometrical and other clinical parameters | 12 weeks
  Improvement of anthropometrical and other clinical parameters during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Hernández Morante, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galindo Munoz JS, Gomez Gallego M, Diaz Soler I, Barbera Ortega MC, Martinez Caceres CM, Hernandez Morante JJ. Effect of a chronotype-adjusted diet on weight loss effectiveness: A randomized clinical trial. Clin Nutr. 2020 Apr;39(4):1041-1048. doi: 10.1016/j.clnu.2019.05.012. Epub 2019 May 21. PMID 31153674